CLINICAL TRIAL: NCT00718341
Title: A Multi-centre, Randomized, Double-blind, Placebo Controlled, Two-period, Crossover Proof-of-concept Study in Male Patients With Fragile X Syndrome to Assess the Efficacy, Safety and Tolerability of Multiple Oral Doses of AFQ056
Brief Title: Efficacy, Safety and Tolerability of AFQ056 in Fragile X Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAFQ056A2204
Record Dates: First submitted 2008-07-17; First posted 2008-07-18 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2010-05

CONDITIONS: Fragile X Syndrome
Keywords: Fragile X Syndrome, adults, efficacy
MeSH Terms: conditions — Fragile X Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: AF056
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AF056
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
This study will evaluate the safety, tolerability and efficacy of multiple doses of AFQ056 in patients with Fragile X Syndrome. The dose range will be 50 to 150 mg b.i.d. The primary read-out of efficacy is reduction in Aberrant-Behavior Checklist score.

ELIGIBILITY:
Inclusion Criteria:

* Male, non-smoking patients between 18 and 35 years of age (both inclusive).
* Patients with fmr1 full mutation (> 200 CGG repeats)
* Patients with a Clinical Global Impression Severity Score (CGI-S) of > 4 (moderately ill)
* Patients with a score of >20 in the ABC-C scale (at screening)
* Patients with a mental age of ≥ 48 months as measured by the Stanford-Binet test

Exclusion Criteria:

* Patients with DSM-IV diagnosis of schizophrenia, history and/or presence of psychosis, confusional states and/or repeated hallucinations.
* Patients with a history of seizures in the past 5 years without any therapeutic treatment controlling the disorders.
* Patients under stable anti-convulsant therapies that experienced seizures in the 2 years prior to randomization
* Patients with ECG abnormalities, autonomic dysfunctions, bronchospastic diseases, drug or atopic allergy
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs
* Patients using (or have used within four weeks before randomization) concomitant medications that are potent inhibitors of CYP3A4 (e.g., ketoconazole, ritonavir, etc.)

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Aberrant-Behavior Checklist- Community Edition

SECONDARY OUTCOMES:
28 days treatment with AFQ056 on behavior (communication, socialization, daily living, repetitive behaviors, anxiety/avoidance, clinical global improvement)
28 days treatment with AFQ056 on cognition (receptive language, attention, vigilance…)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Novartis investigator site
Locations (3):
- Novartis Investigator Site, Bron, France
- Novartis Investigator Site, Rome, Italy
- Novartis Investigator Site, Lausanne, Switzerland

REFERENCES:
- [Derived] Jacquemont S, Curie A, des Portes V, Torrioli MG, Berry-Kravis E, Hagerman RJ, Ramos FJ, Cornish K, He Y, Paulding C, Neri G, Chen F, Hadjikhani N, Martinet D, Meyer J, Beckmann JS, Delange K, Brun A, Bussy G, Gasparini F, Hilse T, Floesser A, Branson J, Bilbe G, Johns D, Gomez-Mancilla B. Epigenetic modification of the FMR1 gene in fragile X syndrome is associated with differential response to the mGluR5 antagonist AFQ056. Sci Transl Med. 2011 Jan 5;3(64):64ra1. doi: 10.1126/scitranslmed.3001708. PMID 21209411